CLINICAL TRIAL: NCT00220064
Title: A Phase II Trial Evaluating Irinotecan With 5_fluorouracil Plus Leucovorin in Patients With Relapsed/Refractory Upper Gastrointestinal Tumours
Brief Title: A Phase II Trial Evaluating Irinotecan Plus 5FU/LV in Patients With Relapsed/Refractory Upper GI Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1810
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Upper Gastrointestinal Tumours
MeSH Terms: interventions — Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irinotecan, 5-Fluorouracil, Leucovorin

SUMMARY:
The objective of this study is to assess the efficacy and toxicity of a 2 weekly regimen containing irinotecan combined with leucovorin-modified 5-fluorouracil in the setting of relapsed or refractory upper gastrointestinal tumours. Patients with locally advanced or metastatic adenocarcinoma originating from the oesophagogastric junction, stomach or pancreas who have previously received chemotherapy and have either failed to respond or who have relapsed after an initial response will be eligible for treatment in this study.

The response rate, failure-free survival and overall survival of treated patients with the two different regimes will be evaluated. Toxicity and quality of life will also be monitored closely.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma or squamous cell carcinoma of the Oesophagus, O-G junction, stomach and pancreas, not amenable to surgical resection.
* Bidimensionally measurable disease, or unidimensional measurable disease accessible by CT scanning, not within previously irradiated areas.
* Patients with progressive disease during previous chemotherapy treatment or within three months of stopping treatment.
* At least one previous chemotherapy regimen, given at least 4 weeks prior to inclusion in this study.
* No previous exposure to irinotecan.
* Adequate bone marrow function with platelets >100 X 109/L; WBC > 3 X 109/L; Neutrophils > 1.5 X 109/L at the time of study entry.
* Satisfactory renal function, serum creatinine 135 mol/litre
* Satisfactory liver function:
* In the absence of liver metastases:- Bilirubin < 1.25N (N=upper limit of normal range) Hepatic transaminases < 2.5N Prothrombin time < 1.5N
* In the presence of liver metastases:- Bilirubin < 1.5N Hepatic transaminases < 5N Prothrombin time < 1.5N
* No uncontrolled medical condition
* No previous malignant disease except for non-melanotic skin cancer or in-situ carcinoma of the uterine cervix.
* ECOG performance status of 0, 1 or 2.
* Predicted life expectancy of > 3 months.
* Adequate contraceptive precautions
* Informed written consent

Exclusion Criteria:

* Medical or psychiatric conditions resulting in inability of patient to give written consent.
* ECOG Performance status >2
* Intracerebral metastases or meningeal carcinomatosis
* Unresolved bowel obstruction
* Uncontrolled angina pectoris, heart failure (New York heart classification 3 or 4).
* Pregnancy/lactation
* Previous malignancy other than adequately treated basal cell carcinoma of the skin or cervical carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2000-07; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Disease stabilization rate or tumour marker response

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust